CLINICAL TRIAL: NCT06207643
Title: Conventional Vs. Eversion Carotid Endarterectomy Immediate and Short-Term Outcomes
Brief Title: Comparison Between Different Techniques for Carotid Artery Endarterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Kariem Ayman Mohamed, assistant lecturer of vascular surgery Sohag university, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-12-01MD
Record Dates: First submitted 2023-12-31; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Carotid Stenosis; Carotid Atherosclerosis; Carotid Artery Plaque
Keywords: carotid endarterectomy
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (A) conventional CEA (Active Comparator): this group of patients will be subjected to carotid endarterectomy using the conventional technique of this procedure
  Interventions: Procedure: carotid endarterectomy
- group (B) Eversion CEA (Active Comparator): this group of patients will be subjected to carotid endarterectomy using the Eversion technique of this procedure
  Interventions: Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: carotid endarterectomy — removing carotid artery atheromatous plaque surgically

SUMMARY:
the goal of this interventional study is to compare between the conventional and the Eversion techniques in performing carotid endarterectomy in patients with carotid artery stenosis the main question it aim to answer is which technique is much more safe and effective the participants will have carotid endarterectomy by one of the two techniques the researcher will compare the group subjected to conventional carotid endarterectomy and the group subjected to Eversion carotid endarterectomy to see which technique is more effective and safe

DETAILED DESCRIPTION:
Carotid endarterectomy (CEA) is widely recognized as the gold standard approach for the prevention of major cerebral events in patients with significant carotid stenosis as it is considered as cerebral revascularization. The procedure entails removing the plaque from the common carotid artery (CCA) and internal carotid artery (ICA) to improve blood flow, prevent potential embolic material and therefore restoring proper cerebral blood flow.

Carotid endarterectomy (CEA) has proven to be a safe and durable operation to decrease the risk of stroke in both symptomatic and asymptomatic patients with extracranial carotid artery stenosis. it is recommended for most symptomatic patients with 50%-99% ICA stenosis. It's considered for asymptomatic patients with 60% - 99%.

There are two main techniques of CEA, conventional carotid endarterectomy (C-CEA) and eversion carotid endarterectomy (E-CEA). More often used is conventional carotid endarterectomy (C-CEA) which is consists of a vertical arteriotomy begun on the CCA and continued through the carotid bifurcation into the ICA beyond the full length of the plaque and closure by patch angioplasty.

As regard comparison between (C-CEA) and (E-CEA) Several studies showed that C-CEA and E-CEA are equally effective surgical approaches for extracranial carotid occlusive disease and studies that compared the influence of E-CEA and C-CEA on postoperative results had varied conclusions some studies have reported no difference in restenosis rates while others have reported less restenosis in eversion endarterectomy. more studies are needed to approve such results, Therefore, it remains difficult to choose the optimal endarterectomy technique.

the study will include 40 patients divided into two groups 20 patients for each group, each group will be subjected to one technique to compare safety and efficacy of each one.

ELIGIBILITY:
Inclusion Criteria:

* Patients having carotid artery stenosis with cerebral events (recent stroke).
* Patients having high grade carotid artery stenosis with increasing symptoms.
* Patients underwent previously CEA presented with carotid restenosis.

Exclusion Criteria:

* Non atherosclerotic carotid artery stenosis e.g., vasculitis, collagen vascular diseases and hypoplastic ICA.
* patients with recently thrombosed ICA.
* High carotid bifurcation to the extent makes CEA not accessible in easy or safe way e.g., increased risk of cranial nerve injury.
* acute ischemic stroke within less than 2 weeks before the procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
postoperative immediate and short term complications | 4 weeks postoperative following end of hospital dismiss
  occurrence of cerebrovascular stroke

CONTACTS AND LOCATIONS:
Overall Officials: kariem Mohamed, Principal Investigator — sohag faculty of medicine
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rerkasem A, Orrapin S, Howard DP, Rerkasem K. Carotid endarterectomy for symptomatic carotid stenosis. Cochrane Database Syst Rev. 2020 Sep 12;9(9):CD001081. doi: 10.1002/14651858.CD001081.pub4. PMID 32918282
- [Background] Uno M, Takai H, Yagi K, Matsubara S. Surgical Technique for Carotid Endarterectomy: Current Methods and Problems. Neurol Med Chir (Tokyo). 2020 Sep 15;60(9):419-428. doi: 10.2176/nmc.ra.2020-0111. Epub 2020 Aug 15. PMID 32801277